CLINICAL TRIAL: NCT06215456
Title: Virtual Reality to Reduce Periprocedural Anxiety During Invasive Coronary Angiography: Rationale and Design of the VR InCard Trial
Brief Title: Virtual Reality to Reduce Periprocedural Anxiety During Invasive Coronary Angiography
Acronym: VR InCard
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 114869
Record Dates: First submitted 2023-12-19; First posted 2024-01-22 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2023-12

CONDITIONS: Anxiety; Anxiety State
Keywords: Virtual reality therapy; Procedural anxiety; Invasive coronary angiography; nonpharmacological; Anxiolysis
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will be treated according to local protocol. Unless contra-indicated, patients experiencing moderate to severe anxiety before undergoing ICA may receive preprocedural oxazepam (10 mg, oral) at the day care unit and diazepam (5 mg, intravenous) before arterial puncture at the catheterization room at nurses and physicians discretion. In patients planned for coronary function testing, benzodiazepines are withheld per protocol.
- Virtual Reality therapy (Active Comparator): The VR intervention group will receive two sessions of VRH in addition to standard care. Before starting the first guided session in this study, patients can use VR during the waiting time using SyncVR Relax & Distract (SyncVR Medical, Utrecht, The Netherlands). Subsequently, the first session of VRH is administered at the day-care unit 20 minutes prior to the procedure. After the first session patients is transported to the catheterization room, where the treatment team have the possibility to introduce themselves to the patients. The second session of VRH is administered during arterial access puncture in the catheterization room, starting 5 minutes prior to puncture and terminating when the diagnostic or guiding coronary catheter is in position. The rest of the procedure will be continued without VR.
  Interventions: Device: Virtual reality therapy

INTERVENTIONS:
Device: Virtual reality therapy — VR therapy will be applied using a head mounted display, the PICO G2 4K headset (Barcelona, Spain). For VRD de application'SyncVR Relax & Distract' (SyncVR Medical, Utrecht, The Netherlands) will be used. This application contains a wide range of relaxation games, relaxing 360 videos, and relaxation exercises each with a duration of 5-20 minutes. Patients can choose videos, games, or exercises according to their own preferences. For VRH sessions, the application HypnoVR (Strasbourg, France) will be used. This app contains several hypnotic narratives integrating sequences of controlled breathing, cardiac coherence, and hypnotic suggestions. Each VRH sessions can be personalized through selecting different environments and musical compositions.The first VRH session will be set to last 20 minutes and the second VRH session will be set to the continuous setting.
  Arms: Virtual Reality therapy

SUMMARY:
Introduction Patients undergoing invasive coronary angiography experience anxiety due to various factors. This can lead to physiological and psychological complications, compromising patient comfort and overall procedural outcomes. Benzodiazepines are commonly used to reduce periprocedural anxiety, although the effect is modest. VR is an promising nonpharmacological intervention that can be used to reduce anxiety in patients undergoing an invasive coronary angiography.

Methods and analysis A single-center open-label randomized controlled trial was performed to assess the effectiveness of add-on VR therapy on anxiety in 100 patients undergoing invasive coronary angiography and experiencing anxiety in periprocedural setting. The primary outcome is the NRS anxiety score measured just before obtaining arterial access. Secondary outcomes are physiological measures of anxiety and the State-Trait Anxiety Inventory, Perceived Stress Scale, and IGroup presence questionnaire. The NRS anxiety level and physiological measurements will be taken at five scheduled times between pre procedural, peri and post procedural. The State-Trait Anxiety Inventory and Perceived Stress Scale will be performed prior to coronary angiography and the State-Trait Anxiety Inventory (state form) and the IGroup Presence questionnaire will be performed post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥16 years undergoing elective cardiac catheterisation
* Patient is willing and able to comply with the study protocol
* NRS anxiety score ≥ 4

Exclusion Criteria:

* History of dementia
* Severe hearing/visual impairment not corrected
* Depression or anxiety disorder

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
NRS anxiety | Assessed at established moment right before start op procedure.
  Numeric rating score for anxiety with 0 representing no anxiety and 10 the worst anxiety imaginable.

SECONDARY OUTCOMES:
NRS anxiety | At set moments: t0 baseline, t1 20-25min preprocedural, t2 20min after t1 right before transfer to procedure room, t3 5 minutes before start procedure, t4 during procedure (directly after arterial access), t5 10min after end of procedure
  Numeric rating score for anxiety with 0 representing no anxiety and 10 the worst anxiety
heart rate | At set moments: t0 baseline, t1 20-25min preprocedural, t2 20min after t1 right before transfer to procedure room, t3 5 minutes before start procedure, t4 during procedure (directly after arterial access), t5 10min after end of procedure
blood pressure | At set moments: t0 baseline, t1 20-25min preprocedural, t2 20min after t1 right before transfer to procedure room, t3 5 minutes before start procedure, t4 during procedure (directly after arterial access), t5 10min after end of procedure
  Both systolic and diastolic blood pressure will be measured
heart rate variability | At set moments: t0 baseline, t1 20-25min preprocedural, t2 20min after t1 right before transfer to procedure room, t3 5 minutes before start procedure, t4 during procedure (directly after arterial access), t5 10min after end of procedure
  LF/HF ratio are extracted
heart rate variability | At set moments: t0 baseline, t1 20-25min preprocedural, t2 20min after t1 right before transfer to procedure room, t3 5 minutes before start procedure, t4 during procedure (directly after arterial access), t5 10min after end of procedure
  RMSSD (root mean square of the successive differences) is extracted
heart rate variability | At set moments: t0 baseline, t1 20-25min preprocedural, t2 20min after t1 right before transfer to procedure room, t3 5 minutes before start procedure, t4 during procedure (directly after arterial access), t5 10min after end of procedure
  SDNN (standard deviation of the NN (R-R) intervals) is extracted
respiration rate | At set moments: t0 baseline, t1 20-25min preprocedural, t2 20min after t1 right before transfer to procedure room, t3 5 minutes before start procedure, t4 during procedure (directly after arterial access), t5 10min after end of procedure
STAI-state short form | At t0 baseline and t5 10min after end of procedure
  State-Trait Anxiety Inventory - state section - 6 item. Score range 6-24. Higher score is higher anxiety.
STAI-trait | At t0 baseline
  State-Trait Anxiety Inventory - trait section - 20 item. Score range 20-80. Higher score is higher anxiety.
Perceived stress questionnaire | At t0 baseline
  The PSS gives an indication about the feelings and thoughts during the past month of the patient. Score range 0-40. Higher score means higher perceived stress.
Pain during arterial punction | At t4 during procedure (directly after arterial access)
  Measured using NRS score, with 0 representing no pain and 10 worst pain imaginable
Patient satisfaction | At t5 10min after end of procedure
  Measured using NRS score, with 0 completely dissatisfied and 10 completely satisfied
Cardiologist satisfaction with procedure | At t5 10min after end of procedure
  Measured using NRS score, with 0 completely dissatisfied and 10 completely satisfied
Radial artery spasm yes/no | At t5 10min after end of procedure
  As reported by cardiologist
complexity of procedure | At t5 10min after end of procedure
  Reported by cardiologist in categories: less complex than anticipated - as anticipated - more complex than anticipated.
anxiolytics use | At t2 20 minutes after t1 right before patients transfers to procedure room and t5 10min after end of procedure
  Use of benzodiazepines (yes/no) was registered for each patient
Igroup presence questionnaire | t5 10min after end of procedure
  Assesses the presence in the virtual environment, only taken in intervention group.
Total finished VR sessions | t5 10min after end of procedure
  Only taken in intervention group.
Total duration of VR use | t5 10min after end of procedure
  Only taken in intervention group.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data will be provided upon reasonable request
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Breunissen EHW, Groenveld TD, Garms L, Bonnes JL, van Goor H, Damman P. Virtual reality to reduce periprocedural anxiety during invasive coronary angiography: rationale and design of the VR InCard trial. Open Heart. 2024 Apr 2;11(1):e002628. doi: 10.1136/openhrt-2024-002628. PMID 38569670